CLINICAL TRIAL: NCT01791231
Title: An Open-Label Study to Investigate the Absorption, Metabolism, and Excretion of JNJ-28431754 in Healthy Male Subjects Following a Single Oral Dose Administration of 14C-JNJ-28431754
Brief Title: A Study to Investigate the Absorption, Metabolism, and Excretion of Canagliflozin (JNJ-28431754) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013624; 28431754NAP1006 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2007-004218-15 (EudraCT Number)
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Healthy; Male; Canagliflozin (JNJ-28431754); Radiolabeled 14C-canagliflozin; Absorption; Metabolism; Excretion; Radioactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolabeled 14C-canagliflozin (Experimental): Each volunteer will receive a single dose of radiolabelled 14C-canagliflozin (14C-JNJ-28431754) on Day 1.
  Interventions: Drug: Radiolabelled 14C-canagliflozin (14C-JNJ-28431754)

INTERVENTIONS:
Drug: Radiolabelled 14C-canagliflozin (14C-JNJ-28431754) — A single oral dose of 196 mg radiolabeled 14C-canagliflozin (14C-JNJ-28431754) liquid suspension containing approximately 40 microcurie (1480 kBq) of 14C radioactivity will be administered on Day 1.
  Other Names: 14C-JNJ-28431754

SUMMARY:
The purpose of this study is to investigate the absorption (the way the drug enters the body), metabolism (the way the drug is broken down in the body), and excretion (the way drug leaves the body) of canagliflozin (JNJ-28431754) in healthy male volunteers after a single dose of radiolabeled 14C-canagliflozin (14C-JNJ-28431754). The safety and tolerability of canagliflozin will also be assessed.

DETAILED DESCRIPTION:
This study will be an open label (all volunteers and study staff know the identity of the assigned treatment), single dose, single center study to investigate the absorption, metabolism, and excretion of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus). The study will consist of 3 phases: a screening phase, an open-label treatment phase, and an end-of study (or follow-up) phase. On Day 1, all volunteers will receive a single oral dose of radiolabeled 14C-canagliflozin which contains 196 mg of canagliflozin and approximately 40 microcurie (1480kBq) of radioactivity. The International Commission on Radiological Protection considers this amount of radioactivity to be acceptable for this type of study. The radioactivity allows the amount of canagliflozin and its metabolites (break-down products) to be more precisely measured in blood, plasma, urine, and feces samples, which will be collected from each volunteer. The total duration of the study is approximately 5 weeks (including screening and follow-up); this time will be increased by 6 days in volunteers who have a slower rate of excretion of canagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) (weight [kg]/height [m2]) between 18 and 30 kg/m2
* Non-smoker

Exclusion Criteria:

* Exposure to radiation for professional or medical reasons (except dental x-rays and x-rays of thorax and bone skeleton, excluding spinal column) in the past 12 months
* History of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin (JNJ-28431754) | Up to Day 3
  Plasma concentrations of canagliflozin (JNJ-28431754) will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug).
Urine concentrations of canagliflozin (JNJ-28431754) | Up to Day 14
  Urine concentrations of canagliflozin (JNJ-28431754) will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug).
Total radioactivity of 14C-canagliflozin (14C-JNJ-28431754) excreted in urine | up to Day 14
  The total radioactivity excreted in the urine will be expressed as a percentage of the administered dose of canagliflozin (JNJ-28431754) and will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug).
Total radioactivity of 14C-canagliflozin (14C-JNJ-28431754) excreted in feces | Up to Day 14
  The total radioactivity excreted in the feces will be expressed as a percentage of the administered dose of canagliflozin (JNJ-28431754) and will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug).
Total radioactivity of 14C-canagliflozin (14C-JNJ-28431754) in blood | Up to Day 8
  The total radioactivity in blood will be used to determine pharmacokinetic parameters for canagliflozin (JNJ-28431754) (measurements describing how the body affects the drug).
Total radioactivity of 14C-canagliflozin (14C-JNJ-28431754) in plasma | Up to Day 8
  The total radioactivity in plasma will be used to determine pharmacokinetic parameters for canagliflozin (JNJ-28431754) (measurements describing how the body affects the drug).
Concentrations of canagliflozin (JNJ-28431754) metabolites in plasma | Up to Day 14
  Concentrations of canagliflozin (JNJ-28431754) metabolites in plasma will be used to investigate the metabolism of canagliflozin (the way the drug is broken down in the body).
Concentrations of canagliflozin (JNJ-28431754) metabolites in urine | Up to Day 14
  Concentrations of canagliflozin (JNJ-28431754) metabolites in urine will be used to investigate the metabolism of canagliflozin (the way the drug is broken down in the body).
Concentrations of canagliflozin (JNJ-28431754) metabolites in feces | Up to Day 14
  Concentrations of canagliflozin (JNJ-28431754) metabolites in feces will be used to investigate the metabolism of canagliflozin (the way the drug is broken down in the body).

SECONDARY OUTCOMES:
Number of volunteers with adverse events as a measure of safety and tolerability | up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium

REFERENCES:
- See also: An Open-Label Study to Investigate the Absorption, Metabolism, and Excretion of JNJ-28431754 in Healthy Male Subjects Following a Single Oral Dose Administration of 14C-JNJ-28431754 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=2027&filename=CR013624_CSR.pdf